CLINICAL TRIAL: NCT06822556
Title: The Effect of TetraSOD® Supplementation on Oxidative Stress Biomarkers, Metabolism and Endurance Exercise Performance in Healthy Adult Males
Brief Title: TetraSOD® Supplementation and Skeletal Muscle Redox Gene Expression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: Fitoplancton Marino, S.L. (Industry)
Responsible Party: Principal Investigator, Stephen Bailey, Dr, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2021-6116-5434
Record Dates: First submitted 2024-12-31; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-12

CONDITIONS: Placebo; Tetraselmis Chuii

STUDY DESIGN:
Intervention Model Description: Crossover Assignment 13 participants completed 2 experimental conditions in a randomized order.
Who Masked: Participant, Investigator
Masking Description: Funder
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo supplementation
  Interventions: Dietary Supplement: Placebo
- Tetraselmis chuii (Active Comparator): Tetraselmis chuii supplementation
  Interventions: Dietary Supplement: Tetraselmis chuii

INTERVENTIONS:
Dietary Supplement: Placebo — 14 days of supplementation with 25 mg/day hemicellulose crystalline
  Arms: Placebo
Dietary Supplement: Tetraselmis chuii — 14 days of supplementation with 25 mg/day tetraselmis chuii
  Arms: Tetraselmis chuii

SUMMARY:
Tetraselmis chuii (TetraSOD) is a marine microalgae that has been reported to improve antioxidant responses in human skeletal muscle cells treated with TetraSOD and to improve recovery from muscle damaging exercise in humans supplemented with TetraSOD. However, the effects of TetraSOD supplementation on human skeletal muscle antioxidant gene expression is less clear.

This study assessed the effect of short-term TetraSOD supplementation on human skeletal muscle antioxidant gene expression in healthy adults.

DETAILED DESCRIPTION:
It is well documented that the production of reactive oxygen species (ROS; unstable molecules that react easily with and damage other molecules in a cell) increases in-line with the intensity and duration of exercise . Although increased ROS production during exercise is initially managed by a variety of 'antioxidants', continued ROS production exceeds the capacity of this antioxidant defense system leading to the development of oxidative stress and impaired exercise performance. Therefore, interventions that can lessen exercise-induced oxidative stress have the potential to improve exercise performance. While dietary supplementation with antioxidant vitamins (e.g. vitamin C and E) has this potential, such interventions do not typically improve exercise performance. Therefore, further research is required to investigate the potential for novel nutritional supplements to lessen exercise-induced oxidative stress and to improve exercise performance. Tetraselmis chuii (TetraSOD) is a natural marine microalgae product. Recent preliminary evidence suggests that treating human skeletal muscle cells with TetraSOD can increase the production of antioxidant enzymes to limit oxidative stress development. In addition, TetraSOD supplementation has been reported to improve recovery from muscle damaging exercise. However, the effects of TetraSOD supplementation on on human skeletal muscle antioxidant gene expression is less clear.

This study assessed the effect of short-term TetraSOD supplementation on human skeletal muscle antioxidant gene expression in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male (as determined by the Health Screening Questionnaire)
* Adult (aged ≥18 and ≤40 years old)
* Recreationally-active (≥2 and ≤4 exercise sessions per week) and a VO2max of ≥ 35 mL/kg/min and ≤ 65 mL/kg/min as determined from the preliminary exercise test
* No known history of gastric, digestive, cardiovascular, renal disease or any other orthopaedic diseases related to motor organs
* Non-smoker
* Healthy body mass index (BMI; ≥18.5 and ≤24.9 kg/m2)
* Not using any dietary supplements, including antioxidant and nitrate-rich supplements, currently or in the past one month
* Not a heavy drinker (≤ 14 units of alcohol) on most weeks
* Not using medication that may affect study measures
* Not participating in other studies currently or in the past two months prior to the consenting session (visit 1) or having an intention to participate in other studies over the period of this study

Exclusion Criteria:

* Female
* Aged <18 and >40 years old
* Sedentary or highly trained with a respective V#O2max of < 35 mL/kg/min and > 65 mL/kg/min as determined from the preliminary exercise test
* History of gastric, digestive, cardiovascular, renal disease or any other orthopaedic diseases related to motor organs
* Smoker
* Unhealthy body mass index (BMI;<18.5 and >24.9 kg/m2)
* Using any dietary supplements, including antioxidant and nitrate-rich supplements, currently or in the past one month
* Heavy drinker (> 14 units of alcohol) on most weeks
* Using medication that may affect study measures
* Participating in other studies currently or in the past two months prior to the consenting session (visit 1) or having an intention to participate in other studies over the period of this study

Participants will be excluded from the biopsy sub-set if they report any of the following:

* Allergy to Lidocaine or any of the ingredients. Symptoms of an allergic reaction may include shortness of breath, wheezing or difficulty breathing, swelling of the face, lips, tongue, or other parts of the body, rash, itching or hives on the skin.
* Infection or swelling where the injection will be given
* Blood infections or disorders
* In severe shock
* Low blood pressure
* Disease of the brain or spinal cord
* Sudden frequent episodes of loss of consciousness
* Myasthenia gravis, a severe muscle weakness
* Heart problems

Furthermore, Lidocaine injection will NOT be used in cases of:

* Severely disturbed cardiac conduction
* Bradycardia
* ADAMS-STOKES syndrome
* Wolfe Parkinson White syndrome
* Sudden heart failure
* Hypersensitivity to amide-type local anaesthetics
* Suspicion of hereditary tendency to malignant hyperthermia
* Disorders of blood coagulation
* Infection of the region to be injected

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Redox and antioxidant gene expression | The primary outcome will be assessed at the end of the 14 day placebo and 14 day Tetraselmis chuii supplementation arms
  112 genes linked to redox and antioxidant responses are expressed as fold-change gene expression (fold-change) determined using the 2-ΔΔCq method.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bailey, Principal Investigator — Loughborough University
Locations (1):
- Loughborough University, Loughborough, United Kingdom, United Kingdom